CLINICAL TRIAL: NCT02717390
Title: Bright by Three (BB3) Effectiveness Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding to recruit target sample size
Sponsor: University of Colorado, Denver (Other)
Collaborators: Bright by 3 (Unknown); Children's Hospital Colorado (Other); Daniels Fund (Unknown); Piton Foundation (Unknown); Gantz Family Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-2164
Record Dates: First submitted 2016-03-15; First posted 2016-03-23 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Developmental Delay
Keywords: Reading; Early Childhood development; Talking; Playing; Praising; Safety; Injury prevention
MeSH Terms: conditions — Learning Disabilities; Speech | interventions — bombesin receptor subtype 3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright By Three (BB3) Intervention (Experimental): The purpose of the BB3 intervention (annual home visit, written materials, and BB3 mobile application 'app') is to increase parental talking, reading, playing, and praise (TRPP) behaviors and improves children's social-emotional and language development at ages 2, 3, and 4 years
  Interventions: Behavioral: Bright By Three (BB3)
- Texts for Child Safety (TCS) Intervention (Active Comparator): The purpose of the injury prevention arm is to reduce the prevalence of safety hazards in the home and car environments, decrease the number of self-reported and medically-attended injuries among children, and increase caregiver's self-reported safety behaviors and knowledge of child safety. The Investigators will compare the results of our tailored child safety intervention (Texts for Child Safety [TCS]) among participants in the injury prevention arm with those randomized to the BB3 arm.
  Interventions: Behavioral: Texts for Child Safety (TCS)

INTERVENTIONS:
Behavioral: Bright By Three (BB3) — The purpose of the BB3 intervention (annual home visit, written materials, and BB3 mobile application 'app') is to increase parental talking, reading, playing, and praise (TRPP) behaviors and improves children's social-emotional and language development at ages 2, 3, and 4 years.
  Arms: Bright By Three (BB3) Intervention
Behavioral: Texts for Child Safety (TCS) — The purpose of the injury prevention arm is to reduce the prevalence of safety hazards in the home and car environments, decrease the number of self-reported and medically-attended injuries among children, and increase caregiver's self-reported safety behaviors and knowledge of child safety. The Investigators will compare the results of our tailored child safety intervention (Texts for Child Safety [TCS]) among participants in the injury prevention arm with those randomized to the BB3 arm.
  Arms: Texts for Child Safety (TCS) Intervention

SUMMARY:
The Investigators propose to conduct a pragmatic randomized controlled trial of 350 one to four year old children and their caregivers to study the effectiveness of 1) the Bright By Three (BB3) intervention for promoting children's language and socio-emotional development and 2) a modified version of the Safe 'N Sound (SNS) intervention for reducing safety hazards and injuries. The SNS intervention will serve as a control for the BB3 group and vice versa so that all study participants will receive a clinically meaningful intervention. In collaboration with primary care clinics that serve low-income and minority children, the Investigators will recruit and randomize 350 twelve to fifteen month olds and their parents/caregivers to one of the two intervention arms and deliver the interventions over a 2 year period.

ELIGIBILITY:
Inclusion Criteria:

* Low-income (based on insurance status of child being Medicaid or CHIP),
* Lower educational level (less than college level education) parents of 12 to 15 month old children from the Rocky Mountain Youth Clinic and the Child Health Clinic who speak either English or Spanish or both and their 12-15 month old toddlers.

Exclusion Criteria:

* Parents with children born prior to 36 weeks gestation (premature infants)
* Children with chronic conditions known to affect neuro-development, such as trisomy 21, or
* Children who have a positive screen on the Children with Special Health Care Needs screener 57
* Parents who have already participated in the BB3 program
* Parents without access to a smart phone
* Parents who cannot read or converse in either English or Spanish

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Change in parental behavior based on the Stim-Q | Child ages 1, 2, 3 and 4
  The Stim-Q assessment tool is a reliable and valid of the cognitive stimulation provided in the home for children between 5 months and 6 years old. It can be completed by a parent in English or Spanish in about 20 minutes and has been used in several studies of interventions to support early childhood development
Change in children's language development based on the CDI | Child ages 1 and 2.
  The MacArthur-Bates Communicative Development Inventories (CDI)-Words and Gestures, Words and Sentences, and CDI-III forms are norm- referenced measures of children's language development that can be completed by a parent in English or Spanish in about 20 minutes for children 8 through 37 months of age.
Change in children's language development based on the E/ROWPVT-4 | Child age 3.
  The Receptive and Expressive One- Word Picture Vocabulary Tests (E/ROWPVT-4) are norm-referenced assessments used to assess receptive and expressive vocabulary skills in children ages 2 years and older who speak English or Spanish. These tests can be administered in-person by a trained research assistant and each take about 20 minutes to complete. Both the CDI and the E/ROWPVT have been used in studies of interventions for language development.

SECONDARY OUTCOMES:
Parental attitudes, norms, self-efficacy, and intentions toward talking, reading, playing, praising (TRPP) behaviors | Child ages 1, 2 and 3
  Measured by a survey similar to the one used in the pilot study - Survey developed by the study team based on the Theories of Planned Behavior and Social Cognitive Theory using measures on attitudes, norms, self-efficacy and intentions validated from other research as a template.
Parental positive regard for the children measured by the Parenting Stress Index | Child ages 1, 2 and 3
  The Parenting Stress Index has been validated with diverse populations to identify dysfunctional parent-child systems in families with infants to 10 year old children, can be completed by a parent in English or Spanish in about 20 minutes, and has been used in hundreds of studies related to early childhood development
Children's socio-emotional development based on the Child Behavior Checklist | Child ages 2 and 3
  The Child Behavior Checklist, Preschool is a validated, commonly used, parent completed tool to identify children ages 1.5 to 5 with emotional and behavioral problems

CONTACTS AND LOCATIONS:
Overall Officials: Mandy Allison, MD, MSPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado AMC, Aurora, Colorado, United States

REFERENCES:
- [Derived] Cunningham MA, Gorman C, McNulty MC, Chavez C, Luna-Asturias C, Dixon CA, Bull S, Berman S, Allison MA. Engage, Develop, Learn: a pilot randomized clinical trial to test if a mobile application can enhance home support for early cognitive development among children living in poverty. Mhealth. 2023 Jan 28;9:4. doi: 10.21037/mhealth-22-13. eCollection 2023. PMID 36760785